CLINICAL TRIAL: NCT00967031
Title: A Multicenter Phase II Clinical Trial Assessing the Efficacy of the Combination of Lapatinib and Capecitabine in Patients With Non Pretreated Brain Metastasis From HER2 Positive Breast Cancer
Brief Title: Lapatinib Ditosylate and Capecitabine in Treating Patients With Stage IV Breast Cancer and Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000642631; EU-20940; GEP 02-0801; 2008-001084-10 (EudraCT Number)
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: HER2-positive breast cancer; male breast cancer; stage IV breast cancer; tumors metastatic to brain
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms, Male; Brain Neoplasms | interventions — Capecitabine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib + capecitabine (Experimental): lapatinib 1250mg/day + capecitabine 2000mg/m2/day
  Interventions: Drug: capecitabine; Drug: lapatinib ditosylate; Other: circulating tumor cell analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: capecitabine
Drug: lapatinib ditosylate
Other: circulating tumor cell analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib ditosylate together with capecitabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving lapatinib ditosylate together with capecitabine works in treating patients with stage IV breast cancer and brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the objective response rate by volumetric analysis of brain metastasis as assessed by MRI in patients with HER2-positive stage IV breast cancer treated with lapatinib ditosylate and capecitabine.

Secondary

* To document any toxicity evaluated by NCI CTC v3.0.
* To assess the time to radiotherapy.
* To document the time to disease progression in the central nervous system (CNS) of these patients.
* To evaluate the overall response rate for extra-CNS disease.
* To assess the clinical benefit (complete response, partial response, and stable disease for ≥ 6 months) for both CNS and extra-CNS disease in these patients.

Tertiary

* To evaluate serum proteomics and metabonomics markers as predictors of response.
* To evaluate the predictive value of circulating tumor cells (CTC) on response.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib ditosylate once daily. Patients also receive oral capecitabine twice daily on days 1-14. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * Stage IV disease
* At least 1 measurable CNS lesion ≥ 10 mm on T1-weighted gadolinium-enhanced MRI

  * No single brain metastasis that could be treated by surgery
* HER-2 positive primary tumor as defined as IHC3+ or IHC2+ and FISH-positive
* Hormone receptor status: not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Absolute Neutrophil Count (ANC) ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10g/dL
* Creatinine ≥ 1.5 times upper limit of normal (ULN)
* Albumin ≥ 2.5 g/dL
* Serum bilirubin ≤ 1.5 times ULN (unless due to Gilbert's syndrome)
* ASAT and ALAT ≤ 3 times ULN (≤ 5 times ULN with documented liver metastasis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks before, during, and for 28 days after completion of study treatment (female) or for 1 week after completion of treatment (male)
* Able to swallow and retain oral medication
* Affiliated to a Social Security System
* No known contraindication to MRI
* No prior or active malignancy, unless disease free for ≥ 10 years
* No other concurrent severe and/or uncontrolled medical disease which could compromise study participation, including any of the following:

  * Infection
  * Cardiac disease (e.g., uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within the past year, Left Ventricular EJection Fraction (LVEF) > grade 2)
  * Current active hepatic or biliary disease (except for Gilbert syndrome, asymptomatic gallstones, liver metastasis or stable chronic liver disease per investigator assessment)
  * Renal disease
  * Active gastrointestinal (GI) tract ulceration, malabsorption syndrome, active uncontrolled ulcerative colitis, or disease significantly affecting GI function
  * Severely impaired lung function (e.g., spirometry and diffusion capacity of lung for carbon monoxide (DLCO) ≤ 50% of normal, and O_2 saturation ≤ 88% at rest on room air)
* No known dihydropyrimidine dehydrogenase deficiency
* No significantly altered mental status prohibiting the understanding of the study, or with psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Not deprived of liberty or placed under the authority of a tutor

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior breast cancer treatment (e.g., trastuzumab, chemotherapy, immunotherapy or biological response modifiers, endocrine therapy, or radiotherapy)
* More than 30 days since prior investigational drugs
* More than 14 days since prior and no concurrent strong inhibitors or inducers of the cytochrome P450 isoenzyme 3A4 (CYP3A4) (i.e., clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir)
* No prior whole brain radiotherapy (WBRT) or brain stereotactic radiotherapy
* No prior treatment with capecitabine and/or lapatinib ditosylate
* No prior resection of the stomach or small bowel
* No concurrent systemic treatment or radiation therapy for breast cancer (except corticosteroid, bisphosphonates, or mannitol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate | february 2012

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTC v3.0 | february 2012
Time to radiotherapy | february 2012
Time to disease progression | february 2012
Overall response rate | february 2012
Clinical benefit (complete response, partial response, and stable disease for at least 6 months) | february 2012
Evaluation of serum proteomics and metabonomics markers as predictors of response | may 2012
Evaluation of the predictive value of circulating tumor cells on response | february 2012

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachelot, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

REFERENCES:
- [Derived] Pierga JY, Bidard FC, Cropet C, Tresca P, Dalenc F, Romieu G, Campone M, Mahier Ait-Oukhatar C, Le Rhun E, Goncalves A, Leheurteur M, Domont J, Gutierrez M, Cure H, Ferrero JM, Labbe-Devilliers C, Bachelot T. Circulating tumor cells and brain metastasis outcome in patients with HER2-positive breast cancer: the LANDSCAPE trial. Ann Oncol. 2013 Dec;24(12):2999-3004. doi: 10.1093/annonc/mdt348. Epub 2013 Sep 6. PMID 24013510
- [Derived] Bachelot T, Romieu G, Campone M, Dieras V, Cropet C, Dalenc F, Jimenez M, Le Rhun E, Pierga JY, Goncalves A, Leheurteur M, Domont J, Gutierrez M, Cure H, Ferrero JM, Labbe-Devilliers C. Lapatinib plus capecitabine in patients with previously untreated brain metastases from HER2-positive metastatic breast cancer (LANDSCAPE): a single-group phase 2 study. Lancet Oncol. 2013 Jan;14(1):64-71. doi: 10.1016/S1470-2045(12)70432-1. Epub 2012 Nov 2. PMID 23122784